CLINICAL TRIAL: NCT00392054
Title: First Line Radiofrequency Ablation Versus Antiarrhythmic Drugs for Atrial Fibrillation Treatment: A Multi-center Randomized Trial
Brief Title: First Line Radiofrequency Ablation Versus Antiarrhythmic Drugs for Atrial Fibrillation Treatment (The RAAFT Study)
Acronym: RAAFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USJan13/09CANAug1/06EUJan1/07
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Paroxysmal; Pulmonary Vein Isolation; Ablation Catheter; Anti-arrhythmic Drug Therapy; First Line Therapy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Catheter Ablation (Experimental): Pulmonary vein isolation performed by catheter ablation for the prevention of recurrence of symptomatic atrial fibrillation
  Interventions: Procedure: Pulmonary Vein Isolation performed by Catheter Ablation
- Antiarrhythmic Drug Therapy (Active Comparator): Conventional antiarrythmic drug therapy for the prevention of recurrence of symptomatic atrial fibrillation
  Interventions: Drug: Conventional Antiarrhythmic Drug Therapy

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation performed by Catheter Ablation — Ablation will be done to achieve entrance block into all pulmonary veins.
  Arms: Catheter Ablation
Drug: Conventional Antiarrhythmic Drug Therapy — Anti-Arrhythmic Drugs per ACC/AHA 2006 Guidelines for the Management of Patients with AF
  Arms: Antiarrhythmic Drug Therapy

SUMMARY:
The purpose of this study is to determine whether catheter-based pulmonary vein isolation is superior to antiarrhythmic drugs as first line therapy in patients with symptomatic paroxysmal recurrent atrial fibrillation not previously treated with therapeutic doses of antiarrhythmic drugs.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia encountered in clinical practice and is estimated to affect 2.2 million people in the United States. AF is a major cause of stroke, adversely affects quality of life, and is associated with increased mortality. Despite advances in antiarrhythmic drug therapy, AF continues to be associated with significant morbidity. Although antiarrhythmic drug therapy is currently considered a first-line option, recent data indicate that more than 35% of Patients will have recurrence of AF despite best antiarrhythmic drug (AAD) therapy, and more than 30% of Patients will discontinue the drugs because of adverse reactions. Furthermore, although recent trials have indicated equivalence of rhythm and rate control strategies in some patient populations, 25-35% of Patients with AF who are rate controlled will continue to have activity limiting symptoms. Newer measures to prevent, treat and potentially cure AF are needed. Seminal work by Haissaguerre and replicated by Chen showed that the majority of AF is initiated by ectopic foci found primarily in the pulmonary veins (PV). Experience with the catheter-based Maze technique led to observations that opened the door to effective and practical catheter-based cures for AF. In response to the difficulties of focal ablation, an alternate strategy has been developed that seeks to electrically isolate the Pulmonary Veins from the atrial tissue. Empirical PV isolation targets all of the PV's without regard to the initiation of ectopic beats. The goal is to create entrance block in the PV. Multipolar circular catheters and basket catheters have been developed that facilitate identification of the electrical connections that are present at the junction of the atrium and the PV, and radiofrequency energy is applied in a circumferential fashion until entrance block is achieved. Relative to focal ablation, circumferential PV isolation is simpler to perform, can be completed without inducing AF, has a shorter procedure time, and has a lower incidence of PV stenosis.

Comparison: Patients will have ablation to achieve entrance and/or exit block into all pulmonary veins, compared with patients receiving antiarrhythmic drugs given in accordance with ACC/AHA/ESC 2006 Guidelines for the Management of patients with AF.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and ≤ 75 years old.
2. Symptomatic, recurrent paroxysmal AF lasting > 30 seconds (at least 4 episodes within the prior 6 months). At least one episode must be documented by Holter,12-lead ECG, event monitor or rhythm strip.

Exclusion Criteria:

1. Documented LVEF <40%.
2. Documented left atrial diameter >5.5cm.
3. Moderate to severe LVH (LV wall thickness >1.5cm).
4. Documented valvular disease, coronary heart disease (defined as the presence of >70% stenosis of coronary arteries or documentation of active myocardial ischemia), post-CABG, postoperative cardiac surgery or peripheral artery disease.
5. Documented AF with electrical cardioversion where full therapeutic antiarrhythmic drug therapy after the cardioversion was prescribed.
6. Untreated hypothyroidism or hyperthyroidism. Patients who are euthyroid on thyroid hormone replacement therapy are acceptable.
7. Contraindication for the use of sotalol, dofetilide and 1C antiarrhythmic drugs(liver enzymes and serum creatinine that are outside the upper normal lab values, e.g. > 3 times ULN with 2 abnormal lab values).
8. Previous left heart ablation procedure, either by surgery or by percutaneous catheter, for atrial fibrillation.
9. Current enrollment in another investigational drug or device study.
10. Presence of any other condition that the investigator feels would be problematic or would restrict or limit the participation of the Patient for the entire study period.
11. Absolute contra-indication to the use of heparin and or warfarin.
12. Increase risk of bleeding, current peptic ulceration, proliferative diabetic retinopathy, history of severe systemic bleeding, or other history of bleeding diathesis or coagulopathy.
13. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD).
14. Documented intra-atrial thrombus, tumor, or another abnormality which precludes catheter introduction.
15. Previous use of full therapeutic dose of an antiarrhythmic drug, including amiodarone, propafenone, flecainide, sotalol, quinidine.
16. Pacemaker or Implantable Cardioverter Defibrillator.
17. Women with a positive pregnancy test.
18. Evidence of active cardiac or systemic infection.
19. Medical condition limiting expected survival to less than one year.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Morillo, MD, Principal Investigator — Population Health Research Institute, Hamilton Health Sciences Corporation and McMaster University; Natale Andrea, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (16):
- United States (2):
  - Texas Cardiac Arrhythmia Foundation, Austin, Texas
  - Austin Heart, Austin, Texas
- Canada (8):
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre University Hospital, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Institut Universitaire de Cardiologie et Pneumologie de Québec, Québec
- Czechia (2):
  - Institute for Clinical and Experimental Medicine, Prague, Prague 4
  - Charles University, Prague
- Germany (3):
  - Abteilung Rhythmologie, Bad Krozingen
  - Asklepios Klinik St. Georg, Hamburg
  - University Hospital Eppendorf, Hamburg
- F. Miulli Hospital, Acquaviva delle Fonti, Bari, Italy

REFERENCES:
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] European Heart Rhythm Association; Heart Rhythm Society; Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Zamorano JL; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation). J Am Coll Cardiol. 2006 Aug 15;48(4):854-906. doi: 10.1016/j.jacc.2006.07.009. No abstract available. PMID 16904574
- [Background] Haissaguerre M, Jais P, Shah DC, Gencel L, Pradeau V, Garrigues S, Chouairi S, Hocini M, Le Metayer P, Roudaut R, Clementy J. Right and left atrial radiofrequency catheter therapy of paroxysmal atrial fibrillation. J Cardiovasc Electrophysiol. 1996 Dec;7(12):1132-44. doi: 10.1111/j.1540-8167.1996.tb00492.x. PMID 8985802
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Chen SA, Tai CT, Tsai CF, Hsieh MH, Ding YA, Chang MS. Radiofrequency catheter ablation of atrial fibrillation initiated by pulmonary vein ectopic beats. J Cardiovasc Electrophysiol. 2000 Feb;11(2):218-27. doi: 10.1111/j.1540-8167.2000.tb00324.x. PMID 10709719
- [Background] Haissaguerre M, Jais P, Shah DC, Garrigue S, Takahashi A, Lavergne T, Hocini M, Peng JT, Roudaut R, Clementy J. Electrophysiological end point for catheter ablation of atrial fibrillation initiated from multiple pulmonary venous foci. Circulation. 2000 Mar 28;101(12):1409-17. doi: 10.1161/01.cir.101.12.1409. PMID 10736285
- [Background] Marrouche NF, Dresing T, Cole C, Bash D, Saad E, Balaban K, Pavia SV, Schweikert R, Saliba W, Abdul-Karim A, Pisano E, Fanelli R, Tchou P, Natale A. Circular mapping and ablation of the pulmonary vein for treatment of atrial fibrillation: impact of different catheter technologies. J Am Coll Cardiol. 2002 Aug 7;40(3):464-74. doi: 10.1016/s0735-1097(02)01972-1. PMID 12142112
- [Background] Ng FS, Camm AJ. Catheter ablation of atrial fibrillation. Clin Cardiol. 2002 Aug;25(8):384-94. doi: 10.1002/clc.4950250808. PMID 12173906
- [Background] Oral H, Chugh A, Good E, Igic P, Elmouchi D, Tschopp DR, Reich SS, Bogun F, Pelosi F Jr, Morady F. Randomized comparison of encircling and nonencircling left atrial ablation for chronic atrial fibrillation. Heart Rhythm. 2005 Nov;2(11):1165-72. doi: 10.1016/j.hrthm.2005.08.003. PMID 16253904
- [Background] Wazni OM, Marrouche NF, Martin DO, Verma A, Bhargava M, Saliba W, Bash D, Schweikert R, Brachmann J, Gunther J, Gutleben K, Pisano E, Potenza D, Fanelli R, Raviele A, Themistoclakis S, Rossillo A, Bonso A, Natale A. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of symptomatic atrial fibrillation: a randomized trial. JAMA. 2005 Jun 1;293(21):2634-40. doi: 10.1001/jama.293.21.2634. PMID 15928285
- [Background] Scherlag BJ, Yamanashi W, Patel U, Lazzara R, Jackman WM. Autonomically induced conversion of pulmonary vein focal firing into atrial fibrillation. J Am Coll Cardiol. 2005 Jun 7;45(11):1878-86. doi: 10.1016/j.jacc.2005.01.057. PMID 15936622
- [Background] Nademanee K, McKenzie J, Kosar E, Schwab M, Sunsaneewitayakul B, Vasavakul T, Khunnawat C, Ngarmukos T. A new approach for catheter ablation of atrial fibrillation: mapping of the electrophysiologic substrate. J Am Coll Cardiol. 2004 Jun 2;43(11):2044-53. doi: 10.1016/j.jacc.2003.12.054. PMID 15172410
- [Derived] Morillo CA, Verma A, Connolly SJ, Kuck KH, Nair GM, Champagne J, Sterns LD, Beresh H, Healey JS, Natale A; RAAFT-2 Investigators. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of paroxysmal atrial fibrillation (RAAFT-2): a randomized trial. JAMA. 2014 Feb 19;311(7):692-700. doi: 10.1001/jama.2014.467. PMID 24549549
- See also: Population Health Research Institute - The RAAFT Study - Sponsor and Central Coordination — http://www.phri.ca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible consenting patients from 16 sites in Canada and Europe were randomly assigned 1:1 to the Catheter Ablation arm or Antiarrythmic Drug Therapy arm. The randomization schedule was computer generated and stratified by site with variable block size.
Period: Overall Study
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Started | 66 (All participants randomized are included in final analysis) | 61 (All participants randomized are included in final analysis)
Received Allocated Intervention | 65 | 60
Completed | 66 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy | Total
Number analyzed (Participants) | 66 | 61 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 48 | 99
  >=65 years | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.3) | 54.3 (11.7) | 55.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 51 | 45 | 96
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
  Czech Republic | 2 | 2 | 4
  Canada | 41 | 38 | 79
  Germany | 16 | 16 | 32
  Italy | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Atrial Tachyarrhythmia
Description: Recurrence of electrocardiographically documented atrial fibrillation, atrial flutter or atrial tachycardia lasting >30 seconds during Follow-up Period. The follow-up period begins 90 days after randomization (the blanking period during which antiarrhythmic drugs are titrated or catheter ablation is performed).
Time Frame: Assessed during 21 month follow-up period
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Groups:
- Catheter Ablation: First-line treatment with radiofrequency catheter ablation procedure
- Antiarrhythmic Drug Therapy: Standard antiarrhythmic drug therapy
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Number analyzed (Participants) | 66 | 61
Participants | 36 | 44
Statistical Analysis 1: Comparison: Catheter Ablation vs Antiarrhythmic Drug Therapy; Event rates were plotted over time using Kaplan-Meier methodology. Only events occurring after the 90-day treatment period were included in the final analysis. Treatment groups were analyzed on an intention-to-treat basis; Test type: Superiority or Other; p = 0.0016, Regression, Cox — Cox regression analysis, stratified by clinical site, was performed and presented as hazard ratios with 95% confidence intervals and a two-sided p-value testing of less than or equal to 0.05 (two-sided) for the Wald test; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.35 to 0.90]

2. Primary Outcome: Comparison of Proportion of Patients With an Occurrence of Any of a Cluster of Serious Complications in Either Arm
Description: Ablation arm cluster: death, cardiac tamponade, severe PV stenosis>70%, atrioesophageal fistula, thromboembolism, vascular complications (i.e. arterial pseudoaneurysm, arteriovenous fistula and hematoma leading to transfusion), phrenic nerve injury or complete AV block requiring permanent pacemaker implantation.
  Antiarrhythmic drug arm cluster: Death, torsade de pointes, bradycardia leading to pacemaker insertion, syncope, QRS duration prolongation > 50% of baseline, 1:1 atrial flutter or any other significant adverse events that leads to drug discontinuation.
Time Frame: Assessed during entire 24 month study period
Population: All patients treated
Measure: Count of Participants; unit: Participants
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Number analyzed (Participants) | 65 | 61
Participants | 5 | 12

3. Secondary Outcome: Number of Participants With Recurrence of Symptomatic Atrial Tachyarrhythmia
Description: Including only symptomatic episodes of all atrial tachyarrhythmias (atrial fibrillation, atrial flutter and atrial tachycardia). The follow-up period begins 90 days after randomization (the blanking period during which antiarrhythmic drugs are titrated or catheter ablation is performed).
Time Frame: 21 months of follow-up
Population: All patients randomized
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Number analyzed (Participants) | 66 | 61
participants | 31 | 36
Statistical Analysis 1: Comparison: Catheter Ablation vs Antiarrhythmic Drug Therapy; Test type: Superiority or Other; p = 0.03, Regression, Cox; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.33 to 0.95]

4. Secondary Outcome: Number of Participants With Recurrence of Symptomatic Atrial Fibrillation
Description: Including only symptomatic episodes of atrial fibrillation in the outcome measure (excluding asymptomatic events and events adjudicated as atrial flutter or atrial tachycardia). The follow-up period begins 90 days after randomization (the blanking period during which antiarrhythmic drugs are titrated or catheter ablation is performed).
Time Frame: During 21 month follow-up period
Population: All patients randomized
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Number analyzed (Participants) | 66 | 61
participants | 27 | 35
Statistical Analysis 1: Comparison: Catheter Ablation vs Antiarrhythmic Drug Therapy; Test type: Superiority or Other; p = 0.017, Regression, Cox; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.3 to 0.89]

5. Secondary Outcome: Episodes of ANY Recurrence of Atrial Tachyarrhythmia
Description: Including all episodes of symptomatic or asymptomatic atrial fibrillation, atrial flutter and atrial tachycardia. The follow-up period begins 90 days after randomization (the blanking period during which antiarrhythmic drugs are titrated or catheter ablation is performed).
Time Frame: During 21 month follow-up period
Population: All patients randomized
Measure: Number; unit: Episodes
Units Other Than Participants: Number of ECGs Adjudicated
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Number analyzed (Participants) | 66 | 61
Number analyzed (Number of ECGs Adjudicated) | 3234 | 3415
Episodes | 213 | 502
Statistical Analysis 1: Comparison: Catheter Ablation vs Antiarrhythmic Drug Therapy; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.28 to 0.4]

6. Secondary Outcome: Number of Participants With Recurrence of Atrial Tachyarrhythmia Obtained Clinically
Description: Including only events documented by 12 lead ECG, Holter monitoring or rhythm strips but excluding TTM monitoring. The follow-up period begins 90 days after randomization (the blanking period during which antiarrhythmic drugs are titrated or catheter ablation is performed).
Time Frame: During 21 month follow-up period
Population: All patients randomized
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Number analyzed (Participants) | 66 | 61
participants | 16 | 19
Statistical Analysis 1: Comparison: Catheter Ablation vs Antiarrhythmic Drug Therapy; Test type: Superiority or Other; p = 0.66, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.42 to 1.72]

7. Secondary Outcome: Quality of Life EQ5D Index Score
Description: The standard EQ-5D questionnaire is completed by study participants. The EQ-5D Index score is a descriptive system comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Self-reported severity for each dimension is given on a 3 level scale: (1) no problems, (2) some problems or (3) major problems. For example a health state: 11223 means: no problems with mobility (1), no problems with self-care (1), some problems with performing usual activity (2), moderate pain/discomfort (2), and major anxiety/depression (3). Thus there are 243 patterns of health state: 11111 to 33333. Scores are converted to a single weighted index score (utility). The index score is derived by applying a formula as developed by Shaw JW, Johnson JA, Coons SJ. US valuation of the EQ-5D health states: development and testing of the D1 valuation model. Med Care 2005; 43(3): 203-220. The final score has a minimum value of 0 and maximum value of 1 (no problems).
Time Frame: Measured at 12 months after randomization
Population: EQ-5D completed at 12 months
Measure: Median (Inter-Quartile Range); unit: Index score
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Number analyzed (Participants) | 59 | 57
Index score | 1 [0.84 to 1] | 1 [0.83 to 1]

8. Secondary Outcome: Quality of Life EQ-5D Visual Analog Score
Description: The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. The scale measures how good/bad one's own health is today, in one's own opinion. 0 means the worst imaginable state of health; 100 means the best imaginable state of health.
Time Frame: Measured At 12 months after randomization
Population: Participants with EQ5D VAS completed at 12 months after randomization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
Number analyzed (Participants) | 59 | 57
score on a scale | 85 [80 to 90] | 80 [75 to 90]

ADVERSE EVENTS:
Time Frame: Duration of follow-up from randomization until completion of follow-up, up to 24 months after randomization. Assessments occurred at 1, 3, 4, 6, 9, 12, 18 and 24 months.
Description: All SAEs (standard definitions) were reported to the central coordinating center within 24 hours of knowledge of the event. A plan was in place for expedited notification to the FDA of any unanticipated fatal or life-threatening adverse events related to either intervention. No such events occurred during study follow-up.
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Therapy
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/60
Serious Adverse Events (participants affected / at risk) | 6/65 | 2/60
Other Adverse Events (participants affected / at risk) | 21/65 | 19/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Catheter Ablation (N=65) | Antiarrhythmic Drug Therapy (N=60)
Angina pectoris (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Post procedural infection (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Pulmonary tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Catheter Ablation (N=65) | Antiarrhythmic Drug Therapy (N=60)
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 0
Adverse drug reaction (General disorders) | 2 | 2
Bronchitis (Infections and infestations) | 3 | 1
joint injury (Injury, poisoning and procedural complications) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Migraine (Nervous system disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Congenital bladder anomaly (Congenital, familial and genetic disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Sensation of foreign body (General disorders) | 1 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Localized infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
urinary tract infection (Infections and infestations) | 1 | 1
Prostate infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase incrased (Investigations) | 1 | 0
Biopsy liver (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Angiogram normal (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No